CLINICAL TRIAL: NCT06181656
Title: Serologic Response to Pneumococcal Vaccination Among Esophageal Cancer Patients With High Grade Lymphopenia After Chemoradiation
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0370; NCI-2023-10646 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Pneumococcal Vaccine; Esophageal Cancer; Lymphopenia; Chemoradiation
MeSH Terms: conditions — Esophageal Neoplasms; Lymphopenia | interventions — SARS-CoV-2 inactivated vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: 30 participants currently receiving, planning to receive, or recently completed chemoradiation for esophageal cancer. This group will be subdivided into Group 1A, which will comprise 15 participants treated with proton therapy, and Group 1B, which will comprise 15 patients treated with intensity modulated radiation therapy (IMRT).
  Interventions: Biological: Pneumonia vaccine
- Group 2: 30 participants currently receiving, planning to receive, or recently completed chemoradiation for hepatocellular carcinoma. This group will be subdivided into Group 2A, which will comprise 15 participants treated with proton therapy, and Group 2B, which will comprise 15 patients treated with intensity modulated radiation therapy (IMRT).
  Interventions: Biological: Pneumonia vaccine
- Group 3: 20 Healthy Volunteers.
  Interventions: Biological: Pneumonia vaccine

INTERVENTIONS:
Biological: Pneumonia vaccine — Given by SC

SUMMARY:
To learn how radiation treatment may affect your responses to vaccines against pneumonia.

DETAILED DESCRIPTION:
Primary Objectives

- Determine the impact of Grade IV radiation-induced lymphopenia on serologic responses to pneumococcal vaccination.

Secondary Objectives

* Determine the impact of chemoradiation on serologic responses to pneumococcal vaccination.
* Determine the impact of radiation modality on serologic responses to pneumococcal vaccination.
* Determine the impact of radiation modality on systemic immunity.
* Determine the incidence of pneumonia among patients treated with a pneumococcal vaccine.
* Determine the impact of radiation modality on pathologic response.
* Determine the impact of radiation modality on intratumoral immunity.
* Determine the relationship between changes in systemic and intratumoral immunity and clinical outcomes (i.e., incidence of pneumonia and pathologic response)
* Determine the impact of tumor histology on serologic responses to pneumococcal vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Group 1A

   a. Patients currently receiving, planning to receive, or recently completed chemoradiation for esophageal cancer with protons.
2. Group 1B

   a. Patients currently receiving, planning to receive, or recently completed chemoradiation for esophageal cancer with intensity-modulated radiation therapy (IMRT)
3. Group 2A

   a. Patients currently receiving, planning to receive, or recently completed definitive proton therapy for unresectable hepatocellular carcinoma.
4. Group 2B

   a. Patients currently receiving, planning to receive, or recently completed definitive IMRT for unresectable hepatocellular carcinoma.
5. Group 3

   a. Healthy age- and gender- matched individuals
6. All Groups

   1. Patients of all genders, races and nationalities will be solicited.
   2. Age >18 years
   3. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with compromised immunologic responses due to an uncontrolled intercurrent immunodeficiency (e.g., Human immunodeficiency virus (HIV), X-linked agammaglobulinemia) or previous or current immune suppressive therapy

  a. Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Patients receiving intravenous immunoglobulin (IVIG) during the study or in the three months prior to study enrollment.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Individuals with previous pneumococcal vaccination in the last 5 years.
* Individuals with severe allergy to any of the vaccine components

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center will enroll 30 esophageal cancer patients. Massachusetts General Hospital in Boston, MA will enroll 30 HCC patients. MD Anderson Cancer Center & Massachusetts General Hospital in Boston will jointly enroll up to 20 health volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Impact of grade IV radiation-induced lymphopenia on serologic responses to pneumococcal vaccination | through study completion; an average of 1 year
  Serologic responses will be calculated as the average fold change in antibody titer for each of 20 pneumococcal serotypes between baseline (time 0) and the first post-vaccination blood draw.

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Lin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org